CLINICAL TRIAL: NCT05838417
Title: Promoting Informed Choice for Breast Cancer Screening: A Longitudinal Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-0957.cc; R37CA254926 (NIH)
Record Dates: First submitted 2023-03-27; First posted 2023-05-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: No known BCRA 1/2 gene mutation; Mammogram; Breast Cancer Screening
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort-1 (Experimental): Individuals who identify as female at birth age 39-49 without a prior breast cancer diagnosis (including DCIS or LCIS) or known BCRA1/2 gene mutations.
  Interventions: Behavioral: REDS survey

INTERVENTIONS:
Behavioral: REDS survey — R - Reactance, E - self-Exemption, D - Disbelief, S - Source derogation

SUMMARY:
All participants will read a decision aid (DA) communicating evidence about mammography screening benefits and harms. Participants' evaluations of that evidence will be assessed, along with their screening intentions and receipt of screening. Participants will be sent 3 surveys via email and a final brief survey conducted by email or phone. The four surveys will be collected 1) upon enrollment and prior to the primary care appointment; 2) following the primary care appointment; 3) 3 months after enrollment; 4) 1 year after enrollment. The final 2 surveys will offer an increased incentive to increase retention rates.

DETAILED DESCRIPTION:
All participants will read a decision aid (DA) communicating evidence about mammography screening benefits and harms. Participants' evaluations of that evidence will be assessed, along with their screening intentions and receipt of screening. Participants will also be asked to report on whether they talked about mammography screening and the content of the DA with their provider. Participants will be sent 3 surveys via email and a final brief survey conducted by email or phone. The four surveys will be collected 1) upon enrollment and prior to the primary care appointment; 2) following the primary care appointment; 3) 3 months after enrollment; 4) 1 year after enrollment. The final 2 surveys will offer an increased incentive to increase retention rates. Time 1 will be an online survey that addresses Aim 1, assessing participants' evaluations of mammography evidence conveyed in the DA. Time 2 will include repeated measures from Time 1 and additionally assess the following: 1. Whether screening was discussed with the provider. 2. If screening was not discussed, why not (e.g. did not want to, no time, other pressing issues, etc.). 3. If screening was discussed, (a) what content from the DA was discussed (i.e. benefits, false positives, overdiagnosis), (b) overall satisfaction with the discussion, (c) whether the provider offered a screening recommendation, (d) open-ended qualitative response eliciting how the discussion went. 4. Whether discussed the BCS-DA with anyone else (e.g., friends or family). 5. Patient activation. 6. Preferred role in decision-making. 7. Perceived barriers to screening. Finally, participants' information environment will be assessed using questions from Pearlman et al. (1997), 8. information seeking (e.g. to what extent the participant valued opinions from the provider, friends, and family), 9. information sharing and communication (e.g. screening attitudes of friends and family), and 10. perception of self as disseminator of mammography-related information. Time 3 will repeat the summary of mammography evidence and measures from Time 2. At Time 4 the team will assess whether screening was received up to one year after study enrollment using the participants' self reports and electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who identify as female at birth
* Ages 39-49 years old (inclusive) at the time of consent
* English literacy
* Internet access
* No prior diagnosis of breast cancer, ductal carcinoma in situ (DCIS, also known as "stage zero breast cancer"), or lobular carcinoma in situ
* No known BCRA1/2 gene mutation

Exclusion Criteria:

* Individuals who identify other than female at birth
* Individuals who are currently pregnant
* Individuals < 39 years old or 50 years old and > at the time of consent
* Lack English literacy
* Lack of internet access
* Prior diagnosis of breast cancer, ductal carcinoma in situ (DCIS, also known as "stage zero breast cancer"), or lobular carcinoma in situ
* Known BCRA1/2 gene mutation
* Decisionally Challenged Individuals
* Prisoners or those on alternative sentencing or probation

Ages: 39 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Identify as female at birth
Enrollment: 700 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
REDS (Reactance, self-Exemption, Disbelief and Source derogation) reactions to mammography benefits | 12 months
  Reactance, self-Exemption, Disbelief and Source derogation in reaction to evidence about mammography benefits. This is a multi-item measure (3-4 questions per subscale) and assessed on a 1 (strongly disagree) to 5 (strongly agree) Likert scale. Averages will be computed to create for scores (corresponding to each sub scale), with a maximum score of 5 and minimum score of 1.
REDS (Reactance, self-Exemption, Disbelief and Source derogation) reactions to mammography harms | 12 months
  Reactance, self-Exemption, Disbelief and Source derogation in reaction to evidence about mammography harms (over diagnosis and false positive results). This is a multi-item measure (3-4 questions per subscale) and assessed on a 1 (strongly disagree) to 5 (strongly agree) Likert scale. Averages will be computed to create for scores (corresponding to each sub scale), with a maximum score of 5 and minimum score of 1. Reactions to over diagnosis and false positives will be assessed separately.
Screening intentions question | 12 months
  This is a single item question in which participants will indicated their intentions to initiate regular screening with mammograms, using a 4 category response: 1. screen now, 2. wait until they are older but before age 50, 3. wait until age 50, or 4. do not intend to screen in the future at any age
Number of participants who receive screening in the study period | 12 months
  We will use medical records to identify whether the participant has received screening in the 12-month study period

SECONDARY OUTCOMES:
Change in breast cancer screening knowledge from pre- to post-decision aid | 12 months
  Breast cancer screening knowledge is assessed immediately before and after the decision aid, and at follow up survey time points. Screening knowledge is assessed with a 10-item multiple choice questionnaire developed in prior research (Hersch et al., 2015). Minimum score=0/10 (0% correct), maximum score=10/10 (100% correct).
Whether the participant had a conversation with their doctor about screening | 12 months
  Assessed after the clinic appointment, participants report whether they talked with their doctor about screening in that appointment using a 3-category response: 1. No, not at all, 2. Yes briefly, 3. Yes in some detail
Change in medical mistrust from pre- to post-decision aid | 12 months
  Medical mistrust (Eaton et al. 2015) is a 6-item validated scale that is administered before the decision aid, after decision aid, and at follow up surveys. Questions are answered using a 1-5 strongly disagree-strongly agree Likert scale. Minimum score=1, maximum score=5.
Perceptions of breast cancer risk | 12 months
  This is a multi-item validated scale to assess perceptions of personal risk, the TRIRISK measure (Ferrer et al. 2016). Scale items are modified to assess perceived breast cancer risk. In this study we assess only the deliberative and affective subscales. Questions are answered using Likert scales. Minimum score=1, maximum score=5.
Emotional responses to the decision aid | 12 months
  The validated Berlin Emotional Responses to Risk Instrument (BERRI; Petrova et al., 2022) is used to assess emotional response to the decision aid. Participants indicate how they felt when they read the decision aid (angry, worried, hopeful, etc.), responding on a 1-7 Likert scale. Mean scores (min=1, max=7) are computed for positive emotion (assured, hopeful, relieved), anxiety (anxious, afraid, worried) and anger (angry, mad).
Whether the participant plans to talk to their doctor about screening in an upcoming appointment | 12 months
  Assessed after the decision aid but before the clinic appointment. Participants indicate whether they intend to discuss breast cancer screening with their doctor using a 4-category response: 1. Definitely not, Probably not, Probably yes, Definitely yes

CONTACTS AND LOCATIONS:
Overall Officials: Laura Scherer, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Hospital, Aurora, Colorado
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No